CLINICAL TRIAL: NCT00706381
Title: Thyroid Hormones Homeostasis and Energy Metabolism Changes During Stimulation of Endogenously Secreted Bile Acids (BAs)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 080165; 08-DK-0165 (Other: NIDDK/NIH)
Record Dates: First submitted 2008-06-26; First posted 2008-06-27 (Estimated); Results first posted 2020-07-22 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2017-08-04

CONDITIONS: Healthy Volunteers
Keywords: Deiodinase; Bile Acids; Cholecystokinin; Thyroid Hormones; Energy Expenditure; Healthy Volunteer
MeSH Terms: interventions — Sincalide; Ursodeoxycholic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- 1: Carb meal, fat meal, sincalide, placebo, urso (Experimental): Participants randomized to consume a 100% carbohydrate meal day 1, then a high fat (72% fat, 8% protein, 20% carbohydrate) meal day 2, IV sincalide 0.04mcg/kg + PO placebo day 3, IV placebo + PO placebo day 4, and IV placebo + PO Ursodiol 15mg/kg day 5
  Interventions: Drug: Sincalide; Drug: Ursodiol; Procedure: Fat Meal; Procedure: Carb meal; Drug: Placebo
- 2: Fat meal, carb meal, sincalide, placebo, urso (Experimental): Participants randomized to consume a high fat (72% fat, 8% protein, 20% carbohydrate) meal day 1, then a 100% carbohydrate meal day 2, IV sincalide 0.04mcg/kg + PO placebo day 3, IV placebo + PO placebo day 4, then IV placebo + PO Ursodiol 15mg/kg day 5
  Interventions: Drug: Sincalide; Drug: Ursodiol; Procedure: Fat Meal; Procedure: Carb meal; Drug: Placebo
- 3: Carb meal, fat meal, placebo, sincalide, urso (Experimental): Participants randomized to consume a 100% carbohydrate meal day 1, then a high fat (72% fat, 8% protein, 20% carbohydrate) meal day 2, IV placebo + PO placebo day 3, IV sincalide 0.04mcg/kg + PO placebo day 4, then IV placebo + PO Ursodiol 15mg/kg day 5
  Interventions: Drug: Sincalide; Drug: Ursodiol; Procedure: Fat Meal; Procedure: Carb meal; Drug: Placebo
- 4: Fat meal, carb meal, placebo, sincalide, urso (Experimental): Participants randomized to consume a high fat (72% fat, 8% protein, 20% carbohydrate) meal day 1, then a 100% carbohydrate meal day 2, IV placebo + PO placebo day 3, IV sincalide 0.04mcg/kg + PO placebo day 4, the IV placebo + PO Ursodiol 15mg/kg day 5
  Interventions: Drug: Sincalide; Drug: Ursodiol; Procedure: Fat Meal; Procedure: Carb meal; Drug: Placebo

INTERVENTIONS:
Drug: Sincalide
Drug: Ursodiol
Procedure: Fat Meal — 600 calorie meal containing 72% fat, 8% protein, and 20% carbohydrate
Procedure: Carb meal — 600 calorie meal containing 100% carbohydrate
Drug: Placebo — IV and/or oral placebo

SUMMARY:
Postprandial thermogenesis, or thermic effect of food are terms that describe the increase in utilization of energy by the human body following a meal. The mechanisms involved in this process are believed to differ according to the type of food consumed, whether fat, protein or carbohydrate.

The bile acids (BAs), unique substances secreted by the gall bladder into the gut after a meal, play an important role in the absorption of fat and the management of cholesterol stores in the body. Recent studies suggest that BAs may also serve as regulators of energy expenditure (consumption) in the cells of our body by increasing the production of T3, an active form of thyroid hormone. T3 in turn is believed to increase the efficiency with which our bodies burn calories thereby generating heat. Although this process has been shown to be effective in rodents who demonstrated weight loss after treatment, the role of BAs in humans is poorly understood. Thus we do not know whether endogenous (produced by the body) or exogenous (taken as medication) BAs play a significant role in the maintenance of body weight. We hypothesize that, similarly to rodents, humans will respond to BAs by increasing energy expenditure via the production of the active form of thyroid hormone.

This randomized, cross-over study will look at changes in thyroid hormones and energy consumption in response to stimuli of endogenous BA secretion including dietary content, and to the intake of pharmacological doses of bile acids.

Following a two-day period of equilibration diet, 30 healthy volunteers will be randomly assigned to receive either a high-fat or high-carbohydrate isocaloric meal followed by a 6-hour metabolic chamber stay; the next day they will be crossed-over to the alternate intervention. During the following three days, the study subjects will again be randomized to receive either an intravenous injection of sincalide (the C-terminal octapeptide fragment of cholecystokinin) 0.04 mcg/kg or placebo and P.O. placebo, or I.V. placebo and 15 mg/kg of BA (ursodiol) with similar metabolic chamber stays and cross-over design.

The data gathered from this study will provide greater insight into the physiological and molecular mechanism(s) regulating the relation between endogenous bile acid secretion and energy metabolism in response to meals, as well as the role of BAs per se on energy metabolism.

DETAILED DESCRIPTION:
Postprandial thermogenesis, or thermic effect of food are terms that describe the increase in utilization of energy by the human body following a meal. The mechanisms involved in this process are believed to differ according to the type of food consumed, whether fat, protein or carbohydrate.

The bile acids (BAs), unique substances secreted by the gall bladder into the gut after a meal, play an important role in the absorption of fat and the management of cholesterol stores in the body. Recent studies suggest that BAs may also serve as regulators of energy expenditure (consumption) in the cells of our body by increasing the production of T3, an active form of thyroid hormone. T3 in turn is believed to increase the efficiency with which our bodies burn calories thereby generating heat. Although this process has been shown to be effective in rodents who demonstrated weight loss after treatment, the role of BAs in humans is poorly understood. Thus we do not know whether endogenous (produced by the body) or exogenous (taken as medication) BAs play a significant role in the maintenance of body weight. We hypothesize that, similarly to rodents, humans will respond to BAs by increasing energy expenditure via the production of the active form of thyroid hormone.

This randomized, cross-over study will look at changes in thyroid hormones and energy consumption in response to stimuli of endogenous BA secretion including dietary content, and to the intake of pharmacological doses of bile acids.

Following a two-day period of equilibration diet, 30 healthy volunteers will be randomly assigned to receive either a high-fat or high-carbohydrate isocaloric meal followed by a 6-hour metabolic chamber stay; the next day they will be crossed-over to the alternate intervention. During the following three days, the study subjects will again be randomized to receive either an intravenous injection of sincalide (the C-terminal octapeptide fragment of cholecystokinin) 0.04 mcg/kg or placebo and P.O. placebo, or I.V. placebo and 15 mg/kg of BA (ursodiol) with similar metabolic chamber stays and cross-over design.

The following parameters will be recorded and compared to placebo:

Energy expenditure

Substrate utilization

Spontaneous movements

Skin and core temperature

Serial changes in circulating thyroid hormones

Serial changes in bile acid serum concentrations

The data gathered from this study will provide greater insight into the physiological and molecular mechanism(s) regulating the relation between endogenous bile acid secretion and energy metabolism in response to meals, as well as the role of BAs per se on energy metabolism.

ELIGIBILITY:
* INCLUSION CRITERIA:

Age greater than or equal to18 years, male or female

Written informed consent

EXCLUSION CRITERIA:

Hypo- or hyperthyroidism (history or serum thyroid-stimulating hormone (TSH) greater than 5.0 or less than 0.4 miU/L)

Blood pressure greater than 140/90 mmHg (26) or receiving antihypertensive therapy

History of cardiovascular disease

BMI less than or equal to 20 or greater than or equal to 27 Kg/m(2)

Diabetes mellitus (fasting serum glucose greater than or equal to 126 mg/dL)

Hyperlipidemia (serum total cholesterol greater than or equal to 240 mg/dL, triglycerides greater than or equal to 220 mg/dL, and/or use of antilipemic therapy)

Liver disease or ALT serum concentrations greater than 1.5 times the upper laboratory reference limit

Hyperbilirubinemia (serum total bilirubin greater than 1.5 mg/dL)

Renal insufficiency or estimated creatinine clearance less than or equal to 50 mL/min (MDRD equation)

Anemia (Hemoglobin concentration less than or equal to 11.1 g/dL females, and 12.7 g/dL males)

History of cholecystectomy or cholelithiasis (by ultrasound at screening).

History of malabsorption, or food allergies/intolerances that would preclude participant from consuming foods required for study

Claustrophobia

History of illicit drug or alcohol abuse within the last 5 years; current use of illicit drugs (by history) or alcohol (CAGE greater than 3)

Psychiatric conditions or behavior that would be incompatible with safe and successful participation in this study

Current use of medications/dietary supplements/alternative therapies known to alter thyroid function, energy expenditure or bile acid secretion

History of weight loss or weight gain of greater than 3 percent body weight over the past 2 months (self-reported)

Pregnancy/breastfeeding/hormonal contraceptive use and childbirth within the last 6 months

Perimenopausal (as self-described within two years from onset of amenorrhea or current complaints of hot flashes)

Current smoker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2008-06-23; Primary Completion 2012-08-21 (Actual); Study Completion 2012-08-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kong Y Chen, Ph.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Hill JO. Understanding and addressing the epidemic of obesity: an energy balance perspective. Endocr Rev. 2006 Dec;27(7):750-61. doi: 10.1210/er.2006-0032. Epub 2006 Nov 22. PMID 17122359
- [Background] Rosen ED, Spiegelman BM. Adipocytes as regulators of energy balance and glucose homeostasis. Nature. 2006 Dec 14;444(7121):847-53. doi: 10.1038/nature05483. PMID 17167472
- [Background] Blaak EE, Hul G, Verdich C, Stich V, Martinez JA, Petersen M, Feskens EF, Patel K, Oppert JM, Barbe P, Toubro S, Polak J, Anderson I, Astrup A, Macdonald I, Langin D, Sorensen T, Saris WH; NUGENOB Consortium. Impaired fat-induced thermogenesis in obese subjects: the NUGENOB study. Obesity (Silver Spring). 2007 Mar;15(3):653-63. doi: 10.1038/oby.2007.606. PMID 17372316
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2008-DK-0165.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 1: Carb Meal, Fat Meal, Sincalide, Placebo, Urso | 2: Fat Meal, Carb Meal, Sincalide, Placebo, Urso | 3: Carb Meal, Fat Meal, Placebo, Sincalide, Urso | 4: Fat Meal, Carb Meal, Placebo, Sincalide, Urso
Started | 10 | 6 | 6 | 9
Intervention 1 (1 Day) | 10 | 6 | 6 | 9
Intervention 2 (1 Day) | 10 | 6 | 6 | 9
Intervention 3 (1 Day) | 10 | 6 | 6 | 9
Intervention 4 (1 Day) | 10 | 5 | 6 | 9
Intervention 5 (1 Day) | 10 | 5 | 5 | 9
Completed | 10 | 5 | 5 | 9
Not Completed | 0 | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- 1: Carb Meal, Fat Meal, Sincalide, Placebo, Urso: Participants randomized to consume a 100% carbohydrate meal day 1, then a high fat (72% fat, 8% protein, 20% carbohydrate) day 2, IV sincalide 0.04mcg/kg + PO placebo day 3, IV placebo + PO placebo day 4, and IV placebo + PO Ursodiol 15mg/kg day 5
- Total: Total of all reporting groups
Arm/Group | 1: Carb Meal, Fat Meal, Sincalide, Placebo, Urso | 2: Fat Meal, Carb Meal, Sincalide, Placebo, Urso | 3: Carb Meal, Fat Meal, Placebo, Sincalide, Urso | 4: Fat Meal, Carb Meal, Placebo, Sincalide, Urso | Total
Number analyzed (Participants) | 10 | 6 | 6 | 9 | 31
Age, Continuous [Mean (Full Range); unit: years] | 30.8 [18 to 55] | 32.3 [20 to 58] | 33.4 [25 to 40] | 30.4 [25 to 40] | 31.6 [18 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 3 | 4 | 15
  Male | 4 | 4 | 3 | 5 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1 | 2
  Not Hispanic or Latino | 8 | 6 | 6 | 7 | 27
  Unknown or Not Reported | 1 | 0 | 0 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 2 | 0 | 6
  White | 5 | 4 | 4 | 7 | 20
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Energy Expenditure
Description: Energy expenditure is measured over 6 hours in a respiratory chamber for each intervention and placebo.
Time Frame: 6 hours
Population: All participants were to participate in all interventions via cross-over design. One patient did not complete the placebo portion and so was eliminated from analysis in all groups. One other participant did not complete the ursodiol portion.
Measure: Mean (Standard Deviation); unit: kcal/min
Groups:
- Carb Meal: All participants who completed the carbohydrate meal and placebo portions of the study
- Fat Meal: All participants who completed the high fat meal and placebo portions of the study
- Sincalide: All participants who completed the sincalide and placebo portions of the study
- Ursodiol: All participants who completed the ursodiol and placebo portions of the study
- Placebo: All participants who completed the sincalide portion of the study
Arm/Group | Carb Meal | Fat Meal | Sincalide | Ursodiol | Placebo
Number analyzed (Participants) | 30 | 30 | 30 | 29 | 30
kcal/min | 1.37 (0.11) | 1.40 (0.09) | 1.28 (0.06) | 1.27 (0.05) | 1.28 (0.05)
Statistical Analysis 1: Comparison: Carb Meal vs Placebo; The percent change from placebo was calculated for each participant and then a t-test was used to test the null hypothesis that this difference was equal to 0; Test type: Superiority; p = 0.0001, t-test, 2 sided; Percent change from placebo = 7.87, Standard Deviation 9.2
Statistical Analysis 2: Comparison: Fat Meal vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, t-test, 2 sided; Percent change from placebo = 9.25, Standard Deviation 8.3
Statistical Analysis 3: Comparison: Sincalide vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.89, Percent change from placebo; Mean Difference (Net) = 0.10, Standard Deviation 6.2
Statistical Analysis 4: Comparison: Ursodiol vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.41, t-test, 2 sided; Percent change from placebo = -0.30, Standard Deviation 7.2

2. Primary Outcome: Bile Acid
Description: Bile acid is measured at 0, 60, 90 and 360 minutes during a 6 hour stay in in a respiratory chamber for each intervention and placebo. The mean of these 4 values is then calculated.
Time Frame: 6 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Placebo: All participants who completed the placebo portion of the study
Arm/Group | Carb Meal | Fat Meal | Sincalide | Ursodiol | Placebo
Number analyzed (Participants) | 30 | 30 | 30 | 29 | 30
mg/dL | 2.89 (0.85) | 7.26 (4.6) | 2.42 (0.64) | 5.17 (1.20) | 2.69 (0.73)
Statistical Analysis 1: Comparison: Carb Meal vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.096, t-test, 2 sided; Percent change from placebo = 40.0, Standard Deviation 72.8
Statistical Analysis 2: Comparison: Fat Meal vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, t-test, 2 sided; Percent change from placebo = 260.4, Standard Deviation 191.7
Statistical Analysis 3: Comparison: Sincalide vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.83, t-test, 2 sided; Percent change from placebo = 16.4, Standard Deviation 56.3
Statistical Analysis 4: Comparison: Ursodiol vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, t-test, 2 sided; Percent change from placebo = 125.7, Standard Deviation 92.2

ADVERSE EVENTS:
Time Frame: 5 days
Groups:
- Carb Meal: All participants who completed the carbohydrate meal portion of the study
- Fat Meall: All participants who completed the high fat meal portion of the study
- Sincalide: All participants who completed the sincalide portion of the study
- Ursodiol: all participants who completed the ursodiol portion of the study
- Placebo: Oral and IV Placebo
Arm/Group | Carb Meal | Fat Meall | Sincalide | Ursodiol | Placebo
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/31 | 0/31 | 0/29 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/31 | 0/31 | 0/29 | 0/30
Other Adverse Events (participants affected / at risk) | 0/31 | 0/31 | 0/31 | 0/29 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-14): https://cdn.clinicaltrials.gov/large-docs/81/NCT00706381/Prot_SAP_000.pdf